CLINICAL TRIAL: NCT01097122
Title: Effects Of Unilateral Forearm Vibration On Electrical Activity Of Untrained Contralateral Forearm Muscle
Brief Title: Effects Of Unilateral Vibration On Contralateral Forearm Muscle Activity
Acronym: BMRR3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vakif Gureba Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ILHAN KARACAN, ILHAN KARACAN, Vakif Gureba Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: VGEAH FTR-3
Record Dates: First submitted 2010-03-27; First posted 2010-04-01 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Osteoporosis; Excitability
Keywords: bone; motor neuron excitability; forearm vibration; mechanical loading; muscle electrical activity
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy young adult subjects (Experimental): Forearm vibration will be applied in healthy young adult subjects
  Interventions: Procedure: Forearm vibration

INTERVENTIONS:
Procedure: Forearm vibration — Mechanical loading with forearm vibration will be applied right radius in all groups
  Other Names: Cyclic mechanical loading

SUMMARY:
This study hypothesize that radius subjecting to mechanical loading may affect excitability of alpha motor neuron innervating muscle, based on its bone mineral density or bone mineral content.

A total of 80 voluntaries are planned to include in this study. Vibration will be applied the right forearm. Muscle electrical activity will be measured on ipsilateral and contralateral flexor carpi radialis (FCR) muscle at rest as EMGrms by surface electromyography (EMG). The rest-EMGrms will be measured at before and during vibration. An increase in muscle electrical activity at rest indicates an increase in motor neuron pool activation. The right distal radius bone mineral content (BMC) and density will be measured by dual energy X-ray absorptiometry (DXA).

The right radius bone mineral density (BMD) and BMC will be evaluated by bone densitometer (GE-LUNAR DPX PRO).

Motor unit potentials will be measured by electromyography at left flexor carpi radialis. Neurotrac ETS device will be used.

DETAILED DESCRIPTION:
A functional cooperation exists between bones and skeletal muscles. Bones work together with muscles as a simple mechanical lever system to produce body movement. One of the important functions of bones is to exert resistance against gravity in order to carry the body. In order to carry out their mechanical functions, bones need to have considerable resistance to deformation under load. It is well-known that muscle activity (i.e., exercises) improves the resistance of bone to mechanical loading, and that it is also important for treating and preventing osteoporosis. Resistance and impact training have been shown to induce bone formation and/or prevent bone resorption. Skeletal muscles have positive effects on bone structure and function. Can bones have an effect on muscle activity? There is only one study about the effect of bones on muscles. In this study, it was shown that bones may affect muscle strength gain in healthy young adult males.

Vibration has a strong osteogenic effect. Vibration-induced bone formation is neuronally regulated. Vibration can also effectively enhance muscle strength and power. Previous studies have shown that vibration increases muscle electromyographic (EMG) activity. But, it has not been reported whether bone has an effect on the increase in muscle EMG activity caused by vibration or not. The aim of this study was to determine whether radius bone exposed to cyclic mechanical loading affects muscle electrical activity of contralateral untrained m. flexor carpi radialis in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Right handed
* Young adult women and men

Exclusion Criteria:

* secondary osteoporosis
* neuropathy (central or peripheral)
* myopathy
* systemic diseases (arthritis, endocrine-metabolic diseases, bone diseases)
* professional sportswoman/sportsman
* subjects doing regular sports activities
* tendinopathy
* amputee, endoprosthesis, metal implants

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Changes in rest muscle electrical activity in the contralateral untrained flexor carpi radialis during the right forearm vibration | 2 or 3 weeks
  Rest muscle electrical activity changes will be examined in the contralateral untrained flexor carpi radialis during the right forearm vibration

CONTACTS AND LOCATIONS:
Overall Officials: ILHAN KARACAN, MD, Study Chair — Vakif Gureba Training & Research Hospital
Locations (1):
- Vakif Gureba Training & Research Hospital, Istanbul, Turkey (Türkiye)